CLINICAL TRIAL: NCT06086691
Title: Effect of Strength Versus Endurance Training on Muscle Damage in Gym Athletes on Caffeine Supplementation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: REC/01241 Mian Waleed Ahmed
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Muscle Damage
Keywords: Caffeine; Creatine Kinase; Endurance Training; Fitness Centers; Skeletal Muscle; Strength Training
MeSH Terms: interventions — Resistance Training; Caffeine; Endurance Training

STUDY DESIGN:
Intervention Model Description: Randomized Crossover Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength Training (Experimental): Strength training exercises along with caffeine supplementation
  Interventions: Other: Strength Training with Caffeine
- Endurance Training (Active Comparator): Endurance training exercises along with caffeine supplementation
  Interventions: Other: Endurance Training with Caffeine

INTERVENTIONS:
Other: Strength Training with Caffeine — The intervention protocol consists of 5 types of strength training exercises. The following exercises will be performed for the strength training group:
  1. bench press (3 sets of 10 reps)
  2. biceps curl (3 sets of 10 reps)
  3. triceps pushdown (3 sets of 10 reps)
  4. leg press (3 sets of 10 reps)
  5. leg extension (3 sets of 10 reps)
  Strength training would be performed in 3 sets of 10 repetitions with 2 minutes of rest between each exercise. This protocol will be performed in a 30-40-minute session. 10-15 minutes of light warm-up activities will be performed before the start of each exercise session. The intervention sessions would be carried out with a 3-5-day gap between the two intervention sessions.
  Arms: Strength Training
Other: Endurance Training with Caffeine — The intervention protocol consists of 3 types of endurance training exercises. The following exercises will be performed by this group:
  1. Cycling (15 min)
  2. Running (20 min)
  3. Rowing (10 min)
  The intervention sessions would be carried out with a 3-5-day gap between the two intervention sessions.
  Arms: Endurance Training

SUMMARY:
Dietary supplements to enhance exercise and athletic performance come in a variety of forms, including tablets, capsules, liquids, powders, and bars. Many of these products contain numerous ingredients in varied combinations and amounts. Among the more common ingredients are amino acids, protein, creatine, and caffeine

DETAILED DESCRIPTION:
Caffeine is a popular nutritional supplement among gym athletes. It is frequently used as an ergogenic aid to improve physical performance, delay fatigue, and increase muscle power. This research aims to evaluate the effectiveness of caffeine through the blood sample test (Serum CK, LDH levels, AST levels) on muscle damage of gym athletes who are performing aerobic and strength training. This study would help understand the effects of strength training and endurance training on muscle damage in gym athletes who are consuming caffeine and to check the serum enzymes level of both groups who are on strength training and those who are on endurance level training, therefore, this study would help determine which athletes should be careful while consuming caffeine for a particular exercise regimen

ELIGIBILITY:
Inclusion Criteria:

* Male gym athletes
* Age: 18-40 years
* Athletes with at least three days training session per week

Exclusion Criteria:

* Athletes already on caffeine supplementation
* Athletes with above normal serum enzyme levels

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Serum CK Levels | Pre-intervention, after 24 hours of the intervention, after 3 days before second intervention, and after 24 hours of the second intervention
  Serum CK level is the amount of an enzyme called creatine kinase (CK) in the blood. CK is a type of protein present in the muscle cells in human body need which is essential for proper functioning. Levels of CK can rise after a heart attack, skeletal muscle injury, or strenuous exercise
Serum LDH levels | Pre-intervention, after 24 hours of the intervention, after 3 days before second intervention, and after 24 hours of the second intervention
  Lactate Dehydrogenase (LDH) is enzyme found in almost every cell of the human body, including your blood, muscles, brain, kidneys, and pancreas.
Serum AST levels | Pre-intervention, after 24 hours of the intervention, after 3 days before second intervention, and after 24 hours of the second intervention
  Aspartate aminotransferase (AST) are enzymes found mainly in the liver, but also found in red blood cells, heart cells, muscle tissue and other organs, such as the pancreas and kidneys.

SECONDARY OUTCOMES:
Rating of fatigue scale/Numeric Rating Scale-Fatigue | Pre-intervention, after 24 hours of the intervention, after 3 days before second intervention, and after 24 hours of the second intervention
  This rating-of-fatigue (ROF) scale has been developed which can track the intensity of perceived fatigue in a variety of contexts.

CONTACTS AND LOCATIONS:
Overall Officials: Noman Sadiq, MS-SPT, Principal Investigator — Riphah International University, Islamabad.
Locations (1):
- Riphah International University (RIU), Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No